CLINICAL TRIAL: NCT02724488
Title: Selection Pressure and Evolution Induced by Immune Checkpoint Inhibitors and Other Immunologic Therapies
Acronym: SPECIAL
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: SPECIAL-001
Record Dates: First submitted 2015-11-19; First posted 2016-03-31 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Melanoma
Keywords: Advanced cancer; Advanced solid tumors; Phase I clinical trial candidates; Phase II clinical trial candidates; Phase III clinical trial candidates; Head and Neck; Melanoma; Upper Aerodigestive cancer; Oral Cavity; Immune Checkpoint Inhibitors; ICIs; ctDNA; Whole Exome Sequencing; Molecular Profiling
MeSH Terms: conditions — Head and Neck Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Part 1: Archival tumor tissue, 3 tubes of whole blood Part 2: Fresh tumor tissue, 5 tubes of whole blood at baseline, serial tubes of whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Part 1: Patients with a histological or cytological diagnosis of advanced solid tumors who are currently on immune checkpoint inhibitors will have archival tumor specimens requested and used for whole exome sequencing (WES) of tumor DNA. 3 tubes of blood at a single time point will be collected for ctDNA analysis and germ line DNA analysis (to study normal variants) using next generation sequencing.
- Part 2: Patients with a histological or cytological diagnosis of advanced solid tumors who are candidates for a phase I, II, or III clinical trial testing immune checkpoint inhibitors (ICIs) or planning to have treatment with ICIs or other immunological therapy as standard of care will have image-guided fresh tumor core needle biopsy at a maximum of 3 time points: 1) prior to commencement of immune checkpoint inhibitors, 2) when disease response to therapy is confirmed using radiology RECIST 1.1 criteria and/or immune related response criteria, and 3) when radiological disease progression is confirmed by using RECIST 1.1. Blood samples for ctDNA analysis will be collected at the commencement of immunotherapy and every 6-12 weeks thereafter until radiological disease progression is confirmed.

SUMMARY:
Two part prospective study to:

1. investigate the feasibility of performing ultra-deep sequencing of plasma derived circulating tumor DNA (ctDNA) in individual patients with advanced solid tumors who are currently being treated with immune checkpoint inhibitors (ICIs) and
2. obtain fresh tumor biopsies and serial blood samples to investigate the clonal evolution of tumors under the selection pressure of ICIs.

DETAILED DESCRIPTION:
This feasibility study will be conducted in two parts.

The first part is mainly designed to investigate the feasibility of performing ultra-deep sequencing of plasma derived circulating tumor DNA (ctDNA) in individual patients with advanced solid tumors who are currently being treated with immune checkpoint inhibitors (ICIs). Patients' archival tumors will be requested and used for whole exome sequencing (WES) of tumor DNA. Blood samples at a single time point will be collected for ctDNA analysis and germ line DNA analysis (to study normal variants) using next generation sequencing.

The second part is designed as a prospective research study in which patients will have tumor and blood samples collected at serial time points to investigate the clonal evolution of tumors under the selection pressure of ICIs. Patients will have image-guided fresh tumor core needle biopsy at a maximum of 3 time points:

1. prior to commencement of ICIs, and
2. when disease response to therapy is confirmed by standard radiology RECIST 1.1 criteria and/or immune related response criteria, and
3. when radiological disease progression on therapy is confirmed by RECIST 1.1 criteria.

Patients who have disease response to immunotherapy could have up to 3 fresh tumor biopsies (all 3 time points) when those who do not respond to therapy will only have one biopsy (1st time point). For patients who will have a mandatory on treatment biopsy as part of a separate clinical trial (within which they are receiving ICIs) at time points different from this study, investigators will request one extra core tumor material for research use within SPECIAL if it is feasible and safe judged by a staff radiologist. Blood samples for ctDNA analysis will be collected at commencement of treatment and every 6-12 weeks thereafter ideally coinciding with radiological tumor assessments whenever possible until radiological disease progression is confirmed using RECIST 1.1 criteria. Normal genomic DNA derived from peripheral mononuclear cells (PBMC) will be extracted from one tube of whole blood collected at baseline to study normal variants. Blood samples for studying changes in immune cells repertoire and immune related amino acids, peptides, proteins and their metabolites in peripheral circulation will be collected at baseline, 6-12 weeks after starting treatment coinciding with the 1st radiological tumor assessment and at the time of radiological disease progression. Imaging parameters for radiomic imaging analysis will be derived from patients' routine CT scans. Fresh tumor biopsies will be used for genomic profiling to study the tumors' mutation spectrum by WES and level of gene expressions. PBMC DNA will be analysed by WES to study normal variants. Mutation profiling of ctDNA will be performed using next generation DNA sequencing approaches.

Genomic data derived from tumor, ctDNA and PBMC DNA analyses will be used to explore tumor clonal architecture and study clonal selection or tumor evolution under selection pressure induced by ICIs or other immunological therapies.

Changes in radiomic imaging signatures during treatment with immune checkpoint inhibitors and their correlation with genomic signatures will also be examined.

Using blood samples collected at baseline, at the time of 1st radiological tumor assessment and at the time of disease progression, dynamic changes in immune cells repertoire and immune related amino acids, peptides, proteins and their metabolites in the peripheral circulation of patients during treatment with ICIs will also be explored.

ELIGIBILITY:
PART 1:

Inclusion Criteria:

1. Age > 18 years.
2. Histological or cytological proof of metastatic solid tumors.
3. Currently receiving immune checkpoint inhibitors or other immunologic therapies of interest (to be determined by study principal investigators).
4. Willingness and ability of patient to provide signed voluntary informed consent.

Exclusion Criteria:

1. Any condition that could interfere with a patient's ability to provide informed consent such as dementia or severe cognitive impairment.
2. Any contraindication to undergoing a venepuncture.

PART 2:

Inclusion Criteria:

1. Age > 18 years.
2. Histological or cytological proof of metastatic solid tumors.
3. At least one biopsiable lesion deemed medically accessible and safe to biopsy.
4. Candidate for one or more phase I or II or III clinical trials with immune checkpoint inhibitors at the time of study enrolment. Patients receiving approved immune checkpoint inhibitors or via special access are also eligible. Patients receiving other immunologic therapies of interest may be allowed (to be determined by study principal investigators).
5. Fulfills local institution's laboratory parameters for tumor biopsy.
6. Willingness and ability of patient to provide signed voluntary informed consent.

Exclusion Criteria:

1. Any condition that could interfere with a patient's ability to provide informed consent such as dementia or severe cognitive impairment.
2. Any contraindication to undergoing a biopsy procedure.
3. Any contraindication to undergoing a venepuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PART 1:
  Patients with a histological or cytological diagnosis of advanced solid tumors who are currently on immune checkpoint inhibitors; fulfill criteria for blood sample collection; and provided written voluntary informed consent.
  PART 2:
  Patients with a histological or cytological diagnosis of advanced solid tumors who are candidates for a phase I, II, or III clinical trial testing immune checkpoint inhibitors or planning to have treatment with ICIs or other immunological therapy as standard of care; have at least one biopsiable lesion deemed accessible and safe to biopsy; fulfill our institution's laboratory parameters for tumor biopsy, and provided written voluntary informed consent.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-04; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: The detection of new mutations from circulating tumor DNA (ctDNA) analyses or change in the frequency of mutations found in archival tumor Whole Exome Sequencing (WES) analyses. | 5 years
Part 2: Concordance between WES analyses of serial tumor biopsies. | 5 years

SECONDARY OUTCOMES:
Part 1: Concordance between DNA analyses of archival tumor and ctDNA analyses. | 5 years
Part 2: Concordance between WES analyses of serial tumor biopsies and ctDNA analyses of serial blood samples. | 5 years
Part 2: Changes in radiomic signatures of tumors between commencement of immune targeted therapies and disease progression assessed from serial CT scans. | 5 years
Part 2: Correlation between tumor radiomic signatures from serial CT scans and genomic profiles (WES and gene expression analyses of serial tumor biopsies and ctDNA samples). | 5 years
Part 2: Changes in levels of immune cells repertoire in peripheral circulation of patients using flow cytometry and related assays. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Hospital, Canada